CLINICAL TRIAL: NCT04436627
Title: Protocol Design of Hand Robotics Assisted Therapy in Patients With Different Severity of Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901693A3
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: Stroke; Robotic Training; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild severity: (Experimental): Brunnstrom stage of distal part: 5-6
  Interventions: Device: Amadeo-assisted training-1
- Moderate severity: (Experimental): Brunnstrom stage of distal part: 4
  Interventions: Device: Amadeo-assisted training-2
- severe severity: (Experimental): Brunnstrom stage of distal part: 2-3
  Interventions: Device: Amadeo-assisted training-3

INTERVENTIONS:
Device: Amadeo-assisted training-1 — Participants will receive 12-15 intervention sessions for about 3 consecutive weeks in a clinical setting (1 hour per session, 4-5 sessions per week). For each intervention session, participants will first receive 20 minutes active assistive training mode, followed by 20 minutes RT functional games (grasp and release) and 20 minutes RT finger coordination training.
  Arms: Mild severity:
Device: Amadeo-assisted training-2 — Participants will receive 12-15 intervention sessions for about 3 consecutive weeks in a clinical setting (1 hour per session, 4-5 sessions per week). For each intervention session, participants will first receive 10 minutes continuous passive motion mode followed by 20 minutes active assistive training mode, and 30 minutes RT functional games (grasp and release).
  Arms: Moderate severity:
Device: Amadeo-assisted training-3 — Participants will receive 12-15 intervention sessions for about 3 consecutive weeks in a clinical setting (1 hour per session, 4-5 sessions per week). For each intervention session, participants will first receive 20 minutes continuous passive motion mode followed by 20 minutes active assistive training mode. After 40 minutes of RT, 20 minutes functional tasks without robot.
  Arms: severe severity:

SUMMARY:
Some studies have shown that the end-effector type of hand robotic-assisted therapy (RT) can effectively improve upper extremity (UE) motor function in patients with stroke. However, these studies provide insufficient information on treatment protocol, making it difficult for therapists to apply the RT in clinical practice. This study aims to develop an end-effector RT treatment protocol and to examine the preliminary effects of the treatment protocol on UE motor function in patients with stroke.

DETAILED DESCRIPTION:
There are two objectives in this case series study. One is combining external scientific evidence with clinical expertise to design a detailed training protocol for RT in patients with different severity of stroke. The other is to examine the effects on UE motor function and explore the client perspective.

The training protocol was developed based on the ACE Star Cycle Knowledge Transformation Model, which includes steps such as summarizing previous evidence and adjusting the protocol after practice by therapists. Purposive sampling will be used to recruit 35patients with stroke with different severities (Brunnstrom stage of distal part: 10 for stage II~III /10 for stage IV /15 for stage V~VI) from a regional hospital in Taiwan. Each participant will receive 12-15 sessions of 50-60 minutes intervention over 3 weeks. Motor function evaluations will be administered before and after the intervention. Wilcoxon Signed Rank test will be used to examine the change between the pretest and posttest.

ELIGIBILITY:
Inclusion Criteria:

* (1) Unilateral stroke patients diagnosed by neurologists with stable life conditions
* (2) Twenty years old or older
* (3) Modified Ashworth Scale of proximal UE ≤ 3 (shoulder and elbow), and Modified Ashworth Scale of distal UE ≤ 2 (wrist and fingers)
* (4) UE subscale of Fugl-Meyer Assessment score < 60
* (5) Cognitive test with the Mini Mental State Examination ≥ 21
* (6) Can provide informed consent

Exclusion Criteria:

* (1) Joint contracture greater than 10° in the paretic wrist or hand
* (2) Absence of proprioception in the wrist and hand
* (3) Other neurological or psychological disorders, e.g. Parkinson's disease
* (4) Receiving Botulinum toxin injections within 3 months
* (5) Enrolling in other rehabilitation experiments or drug studies within 3 months
* (6) unable to operate the AMADEO training system or who may have safety concern

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment, FMA | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The UE subscale of Fugl-Meyer Assessment (UE-FMA) is used to evaluate the recovery of motor function of UE. FMA mainly evaluates the degree of synergy pattern during volitional movements, as well as reflex activity and coordination. UE-FMA consists of 33 items and the total motor score of UE-FMA is 66 points. The higher score means better motor function. FMA has good interrater reliability, good test-retest reliability, and moderate responsiveness.
Modified Ashworth scale of muscle spasticity, MAS | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The Modified Ashworth Scale (MAS) is used to measure muscle spasticity of specific muscle groups of the paretic UE. We measure the muscle tone of proximal part (including shoulder and elbow) and distal part (including wrist and fingers). The grading of spasticity ranges from 0 to 4. A higher score indicates higher levels of spasticity. MAS is a reliable measurement with moderate to high interrater reliability and intrarater reliability.
Grip and pinch power | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The electrical handgrip dynamometers (Jamar® Plus+ Hand Evaluation Kit) is used to assess the strength of hand grasp and lateral pinch (thumb and index) of both hands (distal part of UE). In each time of assessment, the patient grasp the handles in elbow flexion 90° and forearm in neutral position, and then make a maximum but stable power for about 5 seconds. Lateral pinch is assessed in a similar means. Each hand is assessed for three times in turns. Good accuracy (± 1-3%) and good reliability (inter-rater reliability and test-retest reliability) have been demonstrated.
Medical Research Council scale, MRC | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The Medical Research Council scale (MRC) is used to assess muscle strength of the paretic UE. Eight muscle groups (including shoulder flexors, shoulder abductors, elbow flexors, elbow extensors, wrist flexors, wrist extensors, finger MP flexors, and finger MP extensors) is manually tested by the assessor. It is rated in a 6-point ordinal scale, and a higher score indicates stronger muscle.
  MRC has very good inter-rater reliability and intra-rater reliability.
Wolf Motor Function Test, WMFT | Frame: Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The Wolf Motor Function Test (WMFT) is a time-based test that measures UE movements and movement speed during functional tasks. The test includes 15 function-based tasks and 2 strength-based tasks. WMFT has standard template printed on the table to assure the placement of test objects, and the positions of patients in each task are also standardized. The participant is asked to perform the tasks with the affected UE as independently as possible, and as quickly as possible. Two types of scores are recorded during the task: WMFT-TIME (completing time of the task) and WMFT-FAS (functional abilities of the paretic UE). The maximum score of WMFT-TIME is 120 seconds, and a higher score means a slower movement. WMFT-FAS is scored from 0 to 5, and a higher score means a higher level of functional performance, better quality, coordination or precision of paretic UE during the task. WMFT has high interrater reliability, internal consistency, and test-retest reliability.
Nine-hole pegboard test, NPT | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  The Nine-hole pegboard test is used to measure finger dexterity of both UE. The participant is asked to take the pegs from a container (one by one), and place them into the holes on the board. After placing the pegs into nine holes, the participant needs to remove the pegs from the holes back into the container (one by one). All the process needs to be as quickly as possible. The NPT has very good interrater reliability and moderate to high test-retest reliability.
User experience | Baseline, post test immediately after completing 12-15 intervention sessions (around 3 weeks after baseline)
  To understand the experience of using the robot-assisted therapy, a semi-structured interview is conducted to understand the patient's perspective. The interview takes about 10 minutes, recording and verbatim is used for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan